CLINICAL TRIAL: NCT05083780
Title: A Study of Hydroxychloroquine and Chlorphenesin Carbamate in Combination With mFOLFIRINOX in Inoperable Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Hydroxychloroquine and Chlorphenesin Carbamate in Combination With mFOLFIRINOX in Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changhoon Yoo (Other)
Collaborators: Oncocross Co. Ltd. (Industry); CytoGen, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Changhoon Yoo, Associate Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC-201/202-001
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — chlorphenesin carbamate; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mFORFIRINOX, Chlorphenesin Carbamate, Hydroxychloroquine (Experimental)
  Interventions: Drug: Chlorphenesin Carbamate, Hydroxychloroquine

INTERVENTIONS:
Drug: Chlorphenesin Carbamate, Hydroxychloroquine — In addition to the mFOLFIRINOX therapy(backbone therapy), chlorphenesin carbamate 250 mg, and hydroxychloroquine 200 mg will be administered orally twice daily for up to 48 weeks.

SUMMARY:
Pancreatic cancer is the 8th most prevalent cancer in Korea, and its 5-year overall survival rate has shown less than 10% due to its dismal prognosis. To date, the only curative treatment of pancreatic cancer is surgical resection. However, about 60% of patients with pancreatic cancer have been diagnosed as a locally advanced unresectable or metastatic disease at diagnosis owning to its difficulty in the early detection of cancer. The 5-year survival rate has been reported to be less than 25% even with surgical resection. Considering the high rate of metastasis and recurrence, systemic chemotherapy is essential to prolong survival. Therefore, Using AI platforms of RAPTOR (RNA expression-based Anti-symmetrical Pairing Tool for On-demand Response) and ReDRUG (Restoration using the drug for targeting unbalanced gene) developed by Oncocross, Chlorphenesin carbamate, and Hydroxychloroquine were discovered as candidate drugs having anti-metastatic effects.

This study aimed to evaluate the efficacy and safety of hydroxychloroquine and chlorphenesin carbamate in combination with mFOLFIRINOX in patients with inoperable locally advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of age ≥ 19 and < 80 years
2. A patient who meets any of the following criteria at the time of screening or before, and who is scheduled to receive chemotherapy with modified FOLFIRINOX for the first time after screening

   * Locally advanced inoperable pancreatic cancer
   * Metastatic pancreatic cancer
3. One or more measurable lesions by RECIST v 1.1
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 pr 1
5. Estimated life expectancy of at least 12 weeks or more at the discretion of the investigator

Exclusion Criteria:

1. History of major surgery within 4 weeks at the time of screening
2. Symptomatic, uncontrolled brain metastasis or meningeal carcinomatosis
3. History of malignancy within 5 years at the time of screening
4. History of human immunodeficiency virus (HIV) or active hepatitis
5. Active infection requiring systemic antibiotic therapy
6. Patients who have maculopathy or are receiving treatment for corneal or retinal disease, or under follow-up
7. History of acute or subacute intestinal obstruction or paralytic ileus, or a history of chronic diarrhea considered clinically significant at the discretion of the investigator
8. Serious neurological, psychiatric condition including drug abuse or alcoholism, which would prevent the subject from participating in the study
9. Patients with any condition who are considered unsuitable for participation in the study in the judgment of the investigator

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v5.0 | up to 3 years

SECONDARY OUTCOMES:
Rate of Progression-Free Survival | 6, 12 months
Rate of Distant Metastasis-Free Survival | 6, 12 months
Overall Survival | up to 3 years
  Time between study treatment and death
Objective Response Rate | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No